CLINICAL TRIAL: NCT06925568
Title: Clinical Profile, Management Strategies, And Outcome Of Patients With Acute Chest Pain In Regional Referral Hospitals In Tanzania. Protocol For A Prospective, Multi-Centre Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Jakaya Kikwete Cardiac Institute (Other Government)
Responsible Party: Principal Investigator, Chiku Badru Mwimbo, Doctor, Jakaya Kikwete Cardiac Institute
Other Study IDs: AB.123/307/01L/39
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients above 18yrs presenting with acute chest pain or Suspected Acute Coronary Syndrome (ACS).
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational study, so there is no direct intervention. However, the study involves documenting and analyzing the existing management strategies, including
  * use of diagnostic tools ECG, troponin tests, etc
  * Administration of medications such as antiplates and anticoagulants.
  * Reperfusion therapies -thrombolysis, PCI

SUMMARY:
This study aims to understand how patients with acute chest pain are evaluated, treated, and cared for in emergency departments (EDs) at regional hospitals in Tanzania. Chest pain can be caused by many conditions, some of which are life-threatening, like heart attacks (acute coronary syndrome, or ACS). In Tanzania and other low-resource settings, delays in diagnosis and treatment can lead to poor outcomes. This study will document current practices, identify challenges, and link these findings to patient outcomes (e.g., survival, complications) to improve care for future patients.

- Participants: Adults (18 years or older) who come to the ED with chest pain or suspected acute coronary syndrome (heart problem) at the regional referral hospitals in Dar es Salaam, Tanzania. Three regional referral hospitals and one specialized cardiac hospital (Jakaya Kikwete Cardiac Institute) will be involved in this study. Research assistants will collect data during routine care.

During the study, i. Enrollment will take place over 12 months; 317 patients with chest pain will be invited to participate.

ii. Researchers will record:

* How quickly patients receive initial diagnostic tests (e.g., ECG, blood tests for heart damage).
* Treatments given (e.g., medications, procedures to restore blood flow to the heart).
* Patient outcomes over 30 days (e.g., survival, readmission to the hospital, complications like another heart attack or stroke).

iii. Follow-up: Patients will be contacted by phone 30 days after their ED visit to check their health status.

This study is important because-: Chest pain is a common reason for ED visits, but in Tanzania, many patients face delays in diagnosis or lack access to lifesaving treatments. This study will identify gaps in care to help hospitals improve emergency services. Understanding the challenges in chest pain care can empower families to advocate for timely treatment for their loved ones. For Healthcare Providers: The findings will guide hospitals in adopting better protocols (e.g., faster ECGs, improved use of medications) and allocating resources effectively. For Policymakers: Results can inform national strategies to reduce deaths from heart disease in Tanzania.

During the study, participants should know that there will be no changes to care; patients will receive the same care they would normally get. The study only observes and records what happens. Personal information will be kept confidential, and data will be anonymized (no names or identifiers used). Participation is voluntary, and patients can choose to join or refuse without affecting their care.

Key Questions the Study Will Answer

1. How quickly do patients with chest pain get critical tests (like ECGs) and treatments in Tanzanian hospitals?
2. What are the most common barriers to timely care (e.g., lack of equipment, training gaps)?
3. What percentage of patients survive 30 days after a chest pain episode, and what factors influence their outcomes? Potential Benefits

   * Improved Care: Findings may lead to better hospital protocols.
   * Resource Allocation: Highlight where hospitals need more tools (e.g., ECG machines) or medications
   * Global Impact: Lessons from Tanzania can help other low-resource countries improve emergency heart care.

Ethical Considerations

* Approval: The study has been reviewed and approved by ethics committees to ensure patient safety and rights.
* Informed Consent: Participants (or their families, if critically ill) will be asked for permission before joining.

How will results be shared-: Findings will be published in medical journals and shared with Tanzanian hospitals, health officials, and global organizations to drive improvements in emergency care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged eighteen years and above who present at the ED with nontraumatic acute chest pain or suspected acute coronary syndrome and who provided informed consent.

Exclusion Criteria:

1. Patients with known lung cancer.
2. Lost to follow-up
3. The patient arrives in cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nontraumatic patients with acute chest pain or suspected acute coronary syndrome (ACS) presenting to the ED at regional referral hospitals.
Sampling Method: Probability Sample
Enrollment: 317 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 30days

SECONDARY OUTCOMES:
Management provided to ACS patients | 30days
Time intervals taken from the initial hospital presentation to the initial management. | 30days
The occurrence of a major adverse cardiovascular event (MACE) within 30 days after the patient's initial presentation to the emergency department. | 30days
  MACE is defined as any of the following: non-fatal myocardial infarction, urgent revascularization, stroke, cardiac arrest, or cardiogenic shock.
ED readmission within 30 days after the initial visit. | 30days

IPD SHARING:
Plan to Share IPD: No